CLINICAL TRIAL: NCT03997084
Title: Patent Foramen Ovale Closure Reduce in SCUBA-divers
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Joanna Hlebowicz, MD, Associated Professor, Skane University Hospital
Other Study IDs: 2017-01-01
Record Dates: First submitted 2019-06-20; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Patent Foramen Ovale; Decompression Illness
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: phone interviews — phone interviews

SUMMARY:
It has been proposed that there would not be an increased risk of DCI after closure of the interatrial communication, i.e. patent foramen ovale (PFO).

ELIGIBILITY:
Inclusion Criteria:

* catheter-based PFO-closure because of DCI

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all Swedish patients who had had catheter-based PFO-closure
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Dives | 2017-01-01 until 2019-01-01
  Interview based on a questionnaire with questions focusing on the dive habits and DCI events.

IPD SHARING:
Plan to Share IPD: No